CLINICAL TRIAL: NCT02675751
Title: A Prospective Study to Evaluate the Safety and Effectiveness of Wavefront-guided PRK Correction of Myopic Refractive Errors With the iDesign Advanced Wavescan Studio™ System and the Star S4 IR™ Excimer Laser System
Brief Title: Prospective S&E Study of Wavefront-guided PRK for Myopia With iDesign Advanced Wavescan Studio™ System and Star S4 IR™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STAR-115-MIPS
Record Dates: First submitted 2016-02-03; First posted 2016-02-05 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Stable Myopic Refractive Error, With or Without Astigmatism
Keywords: myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- wavefront-guided PRK with iDesign (Experimental): wavefront-guided PRK for treatment of myopic refractive errors based upon measurements obtained with the iDesign System using the STAR S4 IR laser
  Interventions: Device: STAR S4 IR laser with iDesign

INTERVENTIONS:
Device: STAR S4 IR laser with iDesign — Surgeons will perform wavefront-guided PRK for the treatment of myopic refractive errors based upon measurements obtained with the iDesign System using the STAR S4 IR laser.

SUMMARY:
Prospective, multicenter, bilaterally-treated, open-label, non-randomized clinical trial.

ELIGIBILITY:
NOTE: Enrollment open only to military personnel

Inclusion Criteria:

* Signed informed consent and HIPAA authorization.
* Refractive error, based on the iDesign displayed refraction must be myopia with or without astigmatism with sphere up to -8.00 D, and cylinder between 0.00 D and -4.00 D with maximum SE of -10.00 D.
* Anticipated residual stromal bed thickness of at least 250 microns as calculated by the iDesign system.
* Distance Best Spectacle Corrected Visual Acuity (BSCVA) of 20/20 or better
* BSCVA ≥2 lines (≥10 letters) better than distance Uncorrected Visual Acuity (UCVA).
* Less than or equal to 0.75 D difference between cycloplegic and manifest refraction sphere.
* Stable refractive error as defined by a change of ≤1.00 D in MRSE over at least a 12 month time period.
* Any subject eye with a history of contact lens wear within the last 4 weeks must demonstrate refractive stability
* Agreement between manifest refraction (adjusted for optical infinity) and iDesign System refraction chosen for treatment.
* Willing and capable of complying with follow-up examinations for the duration of the study.

Exclusion Criteria:

* Women who are pregnant, breast-feeding, or intend to become pregnant, or not using an adequate method of birth control.
* Concurrent use of systemic (including inhaled) medications that may impair healing.
* History of any of the following medical conditions, or any other condition that could affect wound healing: collagen vascular disease, autoimmune disease, immunodeficiency diseases, ocular herpes zoster or herpes simplex, endocrine disorders (including, but not limited to unstable thyroid disorders and diabetes), lupus, and rheumatoid arthritis.
* Subjects with a cardiac pacemaker, implanted defibrillator or other implanted electronic device.
* History of prior intraocular or corneal surgery, active ophthalmic disease or abnormality, retinal detachment/repair, clinically significant lens opacity, clinical evidence of trauma, corneal opacity within the central 9 mm and visible on topography, at risk for developing strabismus, or with evidence of glaucoma or propensity for narrow angle glaucoma.
* Evidence of keratoconus, corneal dystrophy or irregularity, or abnormal topography
* Known sensitivity or inappropriate responsiveness to any of the medications used in this study.
* If either eye does not meet all inclusion criteria
* Desire to have monovision.
* Participation in any other clinical study, with the exception of the fellow eye in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision Clinical Trials, Study Director — Johnson & Johnson Surgical Vision, Inc.

REFERENCES:
- [Derived] Hofmeister EM, Cason JB, Murdoch DM, Yau IW, Wang Y, Parizadeh DD, Janakiraman DP, Kasthurirangan S. Wavefront-guided PRK treatment of myopia using a refractive aberrometer. J Cataract Refract Surg. 2023 Mar 1;49(3):292-298. doi: 10.1097/j.jcrs.0000000000001083. PMID 36730946

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 235 subjects were consented in the study, of which all 167 subjects have both eyes treated for a total of 334 treated eyes.
Units Other Than Participants: Eyes
Groups:
- PRK Correction With iDesign System and STAR S4 IR Laser: Surgeons performed wavefront-guided PRK for the treatment of myopic refractive errors based upon measurements obtained with the iDesign System using the STAR S4 IR laser
Period: Overall Study
Arm/Group | PRK Correction With iDesign System and STAR S4 IR Laser
Started (Participants 167 Units (eyes) 334) | 167; 334 Eyes
Completed (Participants 151 Units (eyes) 302) | 151; 302 Eyes
Not Completed | 16; 32 Eyes
Not completed — Lost to Follow-up | 16

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Arm/Group | PRK Correction With iDesign System and STAR S4 IR Laser
Number analyzed (Participants) | 167
Number analyzed (Eyes) | 334
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.6 (5.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 114
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 110
  More than one race | 20
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Eyes Achieving the Target of Monocular Uncorrected Visual Acuity of 20/40 or Better
Description: At 6 months, UCVA of 20/40 was achieved in 100% (324/324) of eyes monocularly.
Time Frame: 6 months
Population: Of the 334 eyes (167 subjects) treated in the study, 324 eyes (162 subjects) were available at 6 months for analysis.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | PRK Correction With iDesign System and STAR S4 IR Laser
Number analyzed (Participants) | 162
Number analyzed (Eyes) | 324
Eyes | 324

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | PRK Correction With iDesign System and STAR S4 IR Laser
All-Cause Mortality (participants affected / at risk) | 0/167
Serious Adverse Events (participants affected / at risk) | 10/167
Other Adverse Events (participants affected / at risk) | 0/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRK Correction With iDesign System and STAR S4 IR Laser (N=167)
Retinal Detachment (Eye disorders) | 1 (1)
Anterior Uveitis (Eye disorders) | 1 (1)
Corneal Abrasions (Eye disorders) | 2 (2)
Corneal Infiltrate (Eye disorders) | 2 (2)
Corneal Haze (Eye disorders) | 2 (3)
Corneal Erosion (Eye disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review results communications prior to public release and can embargo communications regarding trial results at any time.

DOCUMENTS (2):
  • Study Protocol (2015-11-17): https://cdn.clinicaltrials.gov/large-docs/51/NCT02675751/Prot_000.pdf
  • Statistical Analysis Plan (2015-11-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT02675751/SAP_001.pdf